CLINICAL TRIAL: NCT00149812
Title: A Clinic-based Program for Families of Depressed Mothers
Brief Title: A Clinic-based Prevention Program for Families of Depressed Mothers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21MH067861 (NIH); R21MH067861 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Depression; Attention Deficit Disorder With Hyperactivity; Conduct Disorder
Keywords: Depression; Child disruptive behavior; Family functioning
MeSH Terms: conditions — Depression; Attention Deficit Disorder with Hyperactivity; Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Intervention: "Keeping Families Strong" Cognitive Behavioral and Communication intervention with mothers recovering from depression and their children, 9 years and older.
  Interventions: Behavioral: Family Functioning Intervention

INTERVENTIONS:
Behavioral: Family Functioning Intervention

SUMMARY:
This study will assess the effectiveness of the "Keeping Families Strong" program (KFS) in avoiding or delaying the onset of psychiatric disorders among children with depressed mothers.

DETAILED DESCRIPTION:
Children of depressed mothers are at high risk for developing serious psychiatric disorders. While genetics can account for about 34% of cases of childhood psychiatric disorders, children of depressed parents are at an even greater risk of developing mental disorders. The "Keeping Families Strong" program, or KFS, was built from evidence-based prevention programs. Its goal is to provide educational, cognitive, and behavioral interventions. These interventions are meant to enhance understanding about depression and its effects on families, improve communication within families, enhance social support, increase positive and consistent parenting, and improve child coping. This will likely improve the children's mental health, as well as positively affect the short- and long-term outcomes of parents recovering from a depressive episode. This study will evaluate the effectiveness of the KFS program in avoiding or delaying the onset of psychiatric disorders among children with depressed mothers.

This 10-week, open-label program will involve 12 meetings, lasting 2 hours each. The parents and the children will attend separate meetings each week on the same nights. Children are prone to take on their parents' responsibilities to prevent them from becoming depressed. In order to avoid this, the children's meetings will focus on clarifying role responsibilities. There will be two additional follow-up meetings in the 3 months following completion of the program. All caregivers are encouraged to participate, including depressed fathers.

ELIGIBILITY:
Inclusion Criteria:

* Parent in treatment for depression
* Parent in maintenance phase of treatment

Exclusion Criteria:

* Active substance abuse
* Substantial cognitive impairment
* Psychosis

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Acceptability of program to parents, children, clinicians, and administrators throughout 10 weeks | 10 weeks

SECONDARY OUTCOMES:
Improvement in the understanding of depression, family communication, parenting practices, and child coping over a one-year period | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anne W. Riley, PhD, Principal Investigator — Bloomberg School of Public Health, Johns Hopkins University
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riley AW, Valdez CR, Barrueco S, Mills C, Beardslee W, Sandler I, Rawal P. Development of a family-based program to reduce risk and promote resilience among families affected by maternal depression: theoretical basis and program description. Clin Child Fam Psychol Rev. 2008 Jun;11(1-2):12-29. doi: 10.1007/s10567-008-0030-3. PMID 18360775
- [Background] Valdez CR, Mills CL, Barrueco S, Leis J, Riley AW. A Pilot Study of a Family-Focused Intervention for Children and Families Affected by Maternal Depression. J Fam Ther. 2011 Feb;33(1):3-19. doi: 10.1111/j.1467-6427.2010.00529.x. PMID 23420650